CLINICAL TRIAL: NCT02266953
Title: The Use of a Communication Tool About Diet in Public Health Nurse Consultations at the Child Health Centre When the Child is Aged 10 Months to 2 Years
Brief Title: The Use of a Communication Tool About Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014/726
Record Dates: First submitted 2014-10-08; First posted 2014-10-17 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2019-12

CONDITIONS: Dietary Intervention
Keywords: Dietary services; Public Health Nursing; Preschool child
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Use of communication tool about diet (Experimental): The children and parents in the intervention group are visiting consultations at the child health centre where the public health nurses use a communication tool about diet in order to promote dialogue about themes concerning food and feeding practices. This intervention is carried out at consultations when the child is 10-, 12- and 15-18 months old.
  Interventions: Behavioral: Use of communication tool about diet
- Treatment as usual (Active Comparator): The children and parents in the control group are visiting consultations at the child health centre where the public health nurses will conduct the consultations as usual and without use of the actual communication tool about diet. The consultations are carried out when the child is 10-, 12- and 15-18 months old.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Use of communication tool about diet — The experimental intervention comprise the public health nurse's use of an image based communication tool in her dialogue with the family. This is in order to act in a patient centered way to facilitate participation by the parents and focus on relevant food and feeding practices from the parents' point of view.
  Arms: Use of communication tool about diet
Behavioral: Treatment as usual — The public health nurses at child health centres in control municipalities are performing consultations at the child health centres as usual and without using the particular communication tool about diet.
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to promote optimal nutrition for the child based on the public health nurse's family-focused conversations at the child health centre. An image based communication tool is used in an intervention in order to promote dialogue and active participation by the parents about themes concerning food and feeding practices.

DETAILED DESCRIPTION:
Norway, as other Nordic countries, has a long-standing tradition of extensive and freely available health care for children under school age at the child health centre. Virtually all parents with small children use these child health centres, having regular encounters with public health nurses. This service aims at promoting health and preventing disease in the population. However, when comes to content and performance of conversation about food and feeding practices there are no guidelines regarding how to adapt the information to the individual child and to his or her family after infancy and up to two years of age.

The overall purpose of this study is to promote optimal nutrition for the child based on the public health nurse's family-focused conversations at the child health centre.

The design of the study is a cluster randomized controlled trial. Statistics Norway has on the basis of a systematic match drawn samples of five pairs of municipalities in Norway. It is random which municipality in each match is extracted respectively to intervention or control municipality.

Public health nurses on child health centres within intervention municipalities will use a communication tool about food and feeding practices in their encounters with participating children and parents when the child is 10-, 12- and 15-18 months old. In the control municipalities corresponding encounters will be as usual, without use of the actual communication tool. The parents will answer a food frequency questionnaire on behalf of their child when the child is 10 months old (baseline) and at the age of two years (final measurement).

Sample size consideration: The aim of the study is to reveal change in vegetable intake. The investigators keep level of statistical significance at the customary 5 % and statistical power of 80 % (beta equal to 20 %), the investigators would need 176 children in each group to reveal the change described above as statistically significant.

The investigators expect some drop out and given that their estimate might be slightly higher, the investigators want to enroll 300 children in each group to make sure our study is sufficiently powered.

Plan for missing data: Concerning missing data the investigators will use mixed models for repeated measure, imputation of missing data will therefore not be necessary. All data will be analysed according to Intention to treat (ITT) analysis.

Analytical principles: Unadjusted (or crude) differences between intervention and control group will be assessed with t-tests (for continuous variables) and Chi-square tests (when we test for association between pairs of categorical data).

In case of continuous outcome variables, the investigators will model the differences between groups (scores from the questionnaires) using uni- and multiple linear regression methods.

All regression models will be conditioned on district variable and not individual level because the randomization was performed on district variable level.

The investigators treat this study as an exploratory analysis, however, they will fit several statistical models and perform several tests therefore a correction for multiple testing will be performed. P-values < 0,01 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. All parents and their children, regardless of the parents' country of origin or native language, who visit the child health centre when the particular child is six months old.
2. Parents that perceive themselves to have sufficient knowledge of Norwegian language to understand the information sheet in Norwegian about the study.

Exclusion Criteria:

1. Parents and their children who do not visit the child health centre when the particular child is six months old.
2. Parents who do not experience to have sufficient knowledge of Norwegian to read and understand the written Norwegian information about the study.
3. The youngest twin and the midst and youngest triplet if the child is a twin or triplet.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 686 (Actual)
Dates: Start 2015-01-05; Primary Completion 2018-06-28 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Increase in the daily intake of vegetables | An expected average of 14 months from baseline
  Metrics are based on parents answering Food Frequency Questionnaires (FFQs) on behalf of their child, at baseline and at endpoint. In addition to questions about the child's diet, there are questions about the child's weight and length at birth, six months, 10 months and 2 years.
  Both FFQs are updated versions, based on validated and standardized FFQs used in earlier national dietary surveys among infants and toddlers in Norway, conducted under the auspices of the University of Oslo, the Norwegian Food Safety Authority and the Norwegian Ministry of Health and Care Services (Spedkost [Infant Diet] 2006-2007 (IS-1635); Småbarnskost [Toddler Diet] 2007 (IS-1731)).
  Analyses of the data will be conducted by use of a diet calculation system. The expectation is an increased intake of 15 g vegetables daily, based on average intake of vegetables of 50 g daily at the age of 1 year according to Spedkost [Infant Diet] 2006-2007 (IS-1635) and Småbarnskost [Toddler Diet]2007 (IS-1731).

SECONDARY OUTCOMES:
Decreased proportion of saturated fat consumed daily | An expected average of 14 months from baseline
  The metrics and analyses are in accordance with those described in the section of primary outcome measure.
  According to the literature, with the intervention the investigators expect a change of 10 % which means the consumption would go down to 10,8 %. Given the small proportions the investigators would need very large numbers of children to reveal such changes as statistically significant. With significance level of 5 % and power of 80 %, they would need 12 426 in each group which is not feasible for us at this stage. Therefore, the secondary aim will be treated as an exploratory analysis and the investigators only aim to describe the proportion of saturated fats consumed daily.

OTHER OUTCOMES:
Change in body weight | An expected average of 14 months from baseline
  The metrics and analysis are in accordance with what is described under the section of primary outcome measure. This outcome measure will be treated as an exploratory analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Glavin, PhD, Study Chair — Oslo Metropolitan University; Sølvi Helseth, Professor, Study Chair — Oslo Metropolitan University
Locations (1):
- Oslo and Akershus University College of Applied Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmberg Fagerlund B, Helseth S, Glavin K. Parental experience of counselling about food and feeding practices at the child health centre: A qualitative study. J Clin Nurs. 2019 May;28(9-10):1653-1663. doi: 10.1111/jocn.14771. Epub 2019 Jan 22. PMID 30618063